CLINICAL TRIAL: NCT03934775
Title: Identification of High-Risk Patients at Admission to an Emergency Department by Non-Invasive Hemodynamics
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Doctor Sofus Carl Emil Friis and Mrs Olga Doris Friss' Fund (Unknown)
Responsible Party: Principal Investigator, Ahmad Sajadieh, Associate professor, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-18062044
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Emergency Department Triage; Non-invasive Hemodynamic
Keywords: emergency department; risk prediction; non-invasive hemodynamic; Heart rate variability
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with acute illness: Patients admitted to the acute medical/emergency department and/or Cardiology department at Bispebjerg Hospital.
  Interventions: Device: Finapres Nova

INTERVENTIONS:
Device: Finapres Nova — Non-invasive mesurement of hemodynamic parameters and heart rate variability

SUMMARY:
The goal of this study is to evaluate the prognostic values of non-invasive hemodynamic parameteres in relation to 30-day mortality and/or acute deterioration in patients who are admitted acutely to the department of emergency medicine or cardiology.

DETAILED DESCRIPTION:
Background

Identification of critically ill and high-risk patients at hospital admission is a major triage task in the emergency department. Rapid identification and treatment of such patients improves survival, reduces complications during admission, duration of hospitalization and the costs of treatment. Reduced heart rate variability (HRV), a marker of autonomic imbalance towards sympathetic dominance, has been shown in several studies to be associated with a poor prognosis in patient groups like myocardial infarction, heart failure, ischemic heart disease, and others. Besides HRV other hemodynamic variables like cardiac stroke volume, cardiac output and peripheral resistance will potentially improve diagnosis of critically ill patients by providing better prognostic value.

Aims & objectives

To develop and validate a prognostic model (based on selected variables derived from Finapres measurements, HRV, CO, and TP) for 30-day mortality and/or acute deterioration in patients who are admitted acutely to the department of emergency medicine or cardiology, University Hospitals of Bispebjerg & Frederiksberg

Methods & Materials

The study is designed as an observational prospective cohort study. The aim is to enroll 1635 patients in total. During a period of 6 to 9 months all patients admitted to the acute medical/emergency department at Bispebjerg Hospital, Copenhagen, Denmark adn who fulfills inclusion criterias will be examined with a 10 minutes examination with the Finapres Nova device. Patients admitted to the departments of medicine/emergency medicine / Cardiology at Bispebjerg Hospital will also be included.

Expected outcomes and perspectives

Several scoring algorithms have been used in the emergency departments to facilitate early recognition of patients with high risk of serious outcomes. There is need to develop better clinical tools to be used in the emergency departments.

The investigators expect to outperform current triage methods by including HRV and hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admittance with acute illness at the department of medicine/emergency medicine / Cardiology at Bispebjerg Hospital
* Able to give informed consent

Exclusion Criteria:

* Terminal disease like advanced cancer or advanced organ failure with a life expectancy of less then three months.
* Candidate for immediate intensive care therapy
* Refuse or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population is patients admitted to the department of emergency medicin and/or cardiology department at Bispebjerg Hospital, Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 942 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
30-day mortality and/or acute deterioration. | 30 days from inclusion
  Death within 30 days and/or cute deterioration in term of unplanned hospital admissions or unplanned transfer to the intensive therapy or any higher level of care.

SECONDARY OUTCOMES:
90-day primary outcome | 90 days from inclusion
  90-day primary outcome
Major Cardiovascular Events (MACE) | 30 days from inclusion
  Composite of cardiovascular death, non-fatal myocardial infarction, coronary revascularization, non-fatal stroke, and hospitalization because of heart failure.
MACE 90-days | 90 days from inclusion
  Composite of cardiovascular death, non-fatal myocardial infarction, coronary revascularization, non-fatal stroke, and hospitalization because of heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Sajadieh, MD, DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malm EHJ, Warrad W, Hadad R, Asmar A, Dominguez H, Haugaard SB, Sajadieh A. Is hyperdynamic circulation a hallmark of obesity? Int J Obes (Lond). 2025 Dec 12. doi: 10.1038/s41366-025-01981-5. Online ahead of print. PMID 41388148